CLINICAL TRIAL: NCT02395640
Title: The Comparison of XELOX and EOX in the First-line Treatment of Advanced Gastric Cancer: An Open-label, Multi-center, Prospective and Randomised Study
Brief Title: The Comparison of XELOX and EOX in the First-line Treatment of Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-EXELOX
Record Dates: First submitted 2015-03-10; First posted 2015-03-23 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2015-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Epirubicin; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- XELOX (Experimental): oxaliplatin 130mg/m2 d1； capecitabine 1000mg/m2 Bid po，d1-14；
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine
- EOX (Active Comparator): Epirubicin 50mg/m2 d1； oxaliplatin 130mg/m2 d1； capecitabine 1000mg/m2 Bid po，d1-14；
  Interventions: Drug: Epirubicin; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Epirubicin — 50mg/m2 ivgtt d1
  Arms: EOX
Drug: Oxaliplatin
  Other Names: 130mg/m2 ivgtt d1
Drug: Capecitabine — 1000mg/m2 po d1-14
  Other Names: Xeloda

SUMMARY:
This study is designed to compare the efficacy and safety of XELOX regimen with EOX regimen in the first-line treatment of advanced gastric cancer patients.

DETAILED DESCRIPTION:
This study is designed to compare the efficacy and safety of XELOX regimen with EOX regimen in the first-line treatment of advanced gastric cancer patients.

ELIGIBILITY:
Major inclusion criteria

* had a histologically proven adenocarcinoma of the gastroesophageal junction, or stomach that was locally advanced (inoperable) or metastatic
* measurable disease, according to the Response Evaluation Criteria in Solid Tumors (RECIST)1.1
* an Eastern Cooperative Oncology Group performance status of 0 to 2
* adequate renal, hepatic, and hematologic function

Major exclusion criteria

* previous chemotherapy or radiotherapy (unless in the adjuvant setting)
* uncontrolled cardiac disease, or other clinically significant, uncontrolled coexisting illness or previous or concurrent cancer
* accumulated dose of Epirubicin exceeds 300mg/m2
* HER2 positive and willing to use trastuzumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2015-03; Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
progression free survival | 7 months

SECONDARY OUTCOMES:
overall survival | 10 months
overall response rate | 2 months
Number of Participants with Adverse Events | 2 months
quality of life questionnaire | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhu XD, Huang MZ, Wang YS, Feng WJ, Chen ZY, He YF, Zhang XW, Liu X, Wang CC, Zhang W, Ying JE, Wu J, Yang L, Qin YR, Luo JF, Zhao XY, Li WH, Zhang Z, Qiu LX, Geng QR, Zou JL, Zhang JY, Zheng H, Song XF, Wu SS, Zhang CY, Gong Z, Liu QQ, Wang XF, Xu Q, Wang Q, Ji JM, Zhao J, Guo WJ. XELOX doublet regimen versus EOX triplet regimen as first-line treatment for advanced gastric cancer: An open-labeled, multicenter, randomized, prospective phase III trial (EXELOX). Cancer Commun (Lond). 2022 Apr;42(4):314-326. doi: 10.1002/cac2.12278. Epub 2022 Feb 25. PMID 35212487